CLINICAL TRIAL: NCT04246528
Title: The Scleroderma Patient-centered Intervention Network (SPIN) Self-Management Program: Protocol for a Randomised Controlled Feasibility Trial With Progression to Full-Scale Trial
Brief Title: SPIN Self-Management Feasibility Trial With Progression to Full-scale Trial (SPIN-SELF)
Acronym: SPIN-SELF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Senior Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-2777
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2023-10

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Scleroderma; Self-management; E-health; Intervention; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Access to the online SPIN-SELF program
  Interventions: Behavioral: SPIN-SELF Program
- Control group (No Intervention): Usual care, no access to the online SPIN-SELF program

INTERVENTIONS:
Behavioral: SPIN-SELF Program — The SPIN-SELF program utilizes social modelling through educational videos of scleroderma patients who describe their own challenges and what they have done to cope with living with scleroderma, as well as videos of patients and health professionals who teach key self-management techniques. The program includes sections on general self-management skills, including goal-setting and self-monitoring), progress tracking, sharing goals and progress with friends and family, and patient stories of experiences with using self-management techniques to cope with SSc symptoms. The program's 9 modules focus on (1) coping with pain; (2) skin care, finger ulcers and Raynaud's; (3) sleep problems; (4) fatigue; (5) gastrointestinal symptoms; (6) itch; (7) managing emotions and stress; (8) coping with body image concerns due to disfigurement; and (9) effective communication with healthcare providers.
  Arms: Intervention group

SUMMARY:
The Scleroderma Patient-centered Intervention Network (SPIN) is an organization established by researchers, health care providers, and people living with scleroderma (systemic sclerosis; SSc) from Canada, the United States, Mexico, Australia, France, Spain, and the United Kingdom. The objectives of SPIN are (1) to assemble a large cohort of SSc patients who complete outcome assessments regularly in order to learn more about important problems faced by people living with SSc and (2) to develop and test a series of internet-based interventions to help patients manage problems related to SSc, including a self-management program (SPIN-SELF Program).

The SPIN-SELF Program was designed by SPIN members based on key tenets of behaviour change that have been successfully incorporated in programs for more common diseases and on patient input. It utilizes social modelling through educational videos of SSc patients describing their challenges and what they have done to cope with SSc, as well as videos teaching key self-management techniques. After an introduction to self-management and instructions on how to navigate the program, patients will have access to modules that are most relevant to their symptoms and disease management challenges. The program's modules address (1) pain; (2) skin care, finger ulcers, and Raynaud's; (3) sleep problems; (4) fatigue; (5) gastrointestinal symptoms; (6) itch; (7) emotions and stress; (8) body image concerns due to disfigurement; and (9) effective communication with healthcare providers.

The proposed study is a feasibility trial with progression to full-scale randomized controlled trial (RCT), depending on whether stoppage criteria are met, of the SPIN Self-Management Program. The SPIN-SELF Program was previously feasibility tested as an online only, self-help intervention. However, uptake was low, thus the investigators have moved to a group-based format. SPIN-SELF participants randomized to intervention will access and use online self-management material, and this will be supported by videoconference group sessions, led by trained peer facilitators.

In the SPIN-SELF feasibility trial with progression to full-scale trial, the investigators will evaluate the disease management self-efficacy of participants who use SPIN-SELF compared to usual care. Eligible SPIN Cohort participants and externally recruited participants, with low disease-management self-efficacy, will be randomized to the SPIN-SELF Program or to usual care only. In the feasibility portion, 40 eligible participants will be randomized. Unless the trial team determines, based on stoppage criteria, that trial procedures need important modifications thereby re-setting the full scale trial as a new trial, the outcome data of the participants in the feasibility portion will be utilized in the analyses of the full-scale trial. In the full-scale RCT, 524 participants will be randomized.

DETAILED DESCRIPTION:
----------------------- OBJECTIVES

The primary objective of the SPIN-SELF feasibility trial with progression to full-scale RCT is to evaluate the disease management self-efficacy of participants who use SPIN's online self-management program (SPIN-SELF), compared to usual care. Secondary objectives are to assess the effect of SPIN-SELF on patient activation (i.e. the extent to which patients effectively engage with and manage their own health), social appearance anxiety, functional health outcomes, as well as usage of the SPIN-SELF program and patient satisfaction with the format and delivery.

----------------------- RECRUITMENT

The SPIN Cohort currently includes over 2000 SSc patients from 47 sites in Canada, the United States, Mexico, Australia, and France, Spain, and the United Kingdom. SPIN Cohort participants complete outcome measures via the Internet upon enrolment and subsequently every three months. Eligible patients, based on questionnaire responses (Self-Efficacy for Managing Chronic Disease (SEMCD) Scale ≤ 7), will be invited to participate in the SPIN-SELF feasibility trial with progression to full-scale trial. Additionally, recruitment announcements for the SPIN-SELF feasibility and full-scale trials will be posted on SPIN's Facebook page and Twitter account and distributed for posting via SPIN's patient organization partners in countries with large English and French-speaking populations. The non-SPIN Cohort participants' eligibility will be assessed with the SEMCD Scale. In the feasibility portion, only English-speaking participants will be included. In the full-scale trial, English and French-speaking participants will be included. An anticipated 40 eligible participants will be recruited into the feasibility portion, and an anticipated 524 eligible participants will be recruited into the SPIN-SELF full-scale RCT.

----------------------- PROGRESSION FROM SPIN-SELF FEASIBILITY TRIAL TO FULL-SCALE TRIAL

The investigators will launch the SPIN-SELF trial as a feasibility trial with possible progression to full-scale trial. Thus, in the feasibility portion of the proposed study, the trial team will collect data to improve several aspects of the trial's processes. At the completion of the feasibility portion, the trial team plans to proceed directly to the full-scale trial, including results from the feasibility stage in the full-scale trial, unless one or more of the stoppage criteria occur. In that case, the trial team will address issues that are identified and begin the full-scale trial anew, separate from the feasibility trial. The stoppage criteria are the following:

1. Recruitment and enrolment of trial participants: If participants who are eligible based on their self-efficacy scores (SEMCD ≤ 7) are not recorded as eligible in the eligibility report on the new SPIN Cohort platform (gen2) and not recruited, then the programming errors in the new platform will need to be addressed and procedures will need to be re-set before the full-scale trial can commence. If more than 6 non-eligible participants (15% of 40 enrolled in feasibility trial) are erroneously identified as eligible and assigned to the intervention or waitlist control, the trial team would address programming errors, modify procedures and conduct the full-scale trial as a new trial.
2. Fidelity of the delivery of the intervention (i.e., group sessions): If by the end of the feasibility trial > 20% of the components of the 8 sessions were not delivered according to the pre-specified program, the trial team will investigate to identify barriers to the delivery of the intervention and will modify the intervention procedures accordingly, before proceeding to the full-scale trial. The full-scale trial would need to commence as a new trial.
3. Group format of the SPIN-SELF sessions: If participants across groups consistently suggest similar changes to the format of the SPIN-SELF program, then the trial team would modify the format of the intervention sessions according to this consensus feedback. These modifications would be made before commencing the full-scale trial as a new trial.

   At the end of the SPIN-SELF feasibility trial, the investigators will use the collected information and evaluation of the stoppage criteria to decide whether to: (1) Continue to the full-scale RCT without modifications to the trial procedures, (2) Modify trial procedures based on participant feedback before continuing to the full-scale trial, or (3) Modify the trial procedures before re-setting them and conducting the full-scale RCT as a new trial (in this case, outcome data collected during the feasibility phase will not be included in the analyses of the full-scale trial).

   ----------------------- RANDOMISATION

   Monthly, consented participants will be entered into pools based on language and scheduling availability. De-identified codes for participants in each pool will be provided to an external randomisation service. Starting with the largest pool, the service will randomly select the largest possible even number of participants (12 to 20 participants) then randomly allocate half to intervention and half to control via single block randomisation using R version 3.6.3. This will be repeated to form as many groups of 6-10 participants and paired waitlist participants as possible each month until the enrolment target is met.

   ----------------------- INTERVENTION

   The SPIN-SELF Program is an 8-session group videoconference intervention that is delivered over the course of 12 weeks. Each videoconference-based intervention group will be led by a facilitator who has been trained in the SPIN- Scleroderma Support Group Leader Education (SSLED) Program.

   ----------------------- STATISTICAL ANALYSES

   Consistent with the feasibility trial design and small sample size, no hypothesis tests are planned for the feasibility portion of the trial. Instead, the investigators will present a description of the feasibility elements, including participants' eligibility and recruitment and numbers and percentages of participants who respond to follow-up measures. Use of the internet intervention will be described by presenting the frequency of logins and usage of the specific SPIN-SELF modules. Analysis of outcome measures will include the completeness of data and presence of floor or ceiling effects. Descriptive statistics will be used to provide means and standard deviations for the measures. Qualitative information on participants' experience using the SPIN-SELF intervention will be used to interpret acceptability related to the group-sessions format, content of the sessions and online program, webpage organization, and navigation. Information related to required resources and management of the program during feasibility will inform any necessary changes to intervention or trial procedures.

   In the full-scale trial, for continuous outcomes, the investigators will use an intent-to-treat analysis to estimate score differences between intervention and waitlist participants with a linear mixed-effects model fit using the lmer function in lme4. Score differences and Hedges' g SMD effect size will be presented with 95% confidence intervals (CIs). To estimate odds ratios for the dichotomous MCID, intent-to-treat analysis will be done with a binomial generalized linear mixed-effects models with a log link function fit using the glmer function in lme4.

   For all models, to account for clustering in the blocked PN-RCT design, the investigators will fit a random intercept and slope for treatment effect by randomisation block and an additional random slope for treatment by intervention group cluster. In main analyses, in addition to a fixed effect for assignment to the intervention arm, the investigators will include a fixed effect for baseline score. In adjusted analyses, the investigators will also control for age (years), sex (male vs. female), SSc disease subtype (diffuse vs. limited), disease duration (years since diagnosis), and country (Canada, France, USA, other) as fixed effects.

   In the event of missing outcome data, to minimize the possibility of bias, the investigators will use multiple imputation by chained equations using the mice package to generate 20 imputed datasets, using 15 cycles per imputed dataset. Variables in the mice procedure will include randomisation block, intervention arm, number of intervention sessions attended, measures of all primary and secondary outcomes at baseline and post-intervention, age, sex, SSc disease subtype, years since diagnosis, country, and race/ethnicity. Pooled standard errors and associated 95% CIs will be estimated using Rubin's rules.

   To estimate average intervention effects among compliers, which will be defined based on the number of sessions completed, the investigators will use an instrumental variable approach to inflate intent-to-treat effects from main models by the inverse probability of compliance among intervention arm participants; 95% CIs will be constructed via a cluster bootstrap approach, resampling at study randomisation block and participant levels. For transparency, results for participants with complete data will also be shown. Participant satisfaction scores for the intervention group will be reported descriptively. All outcome analyses will be conducted in R (R version 3.6.3; R Studio version 1.2.5042). All analyses will be 2-sided with alpha = 0.05. The investigators will not adjust for multiple analyses since a single primary outcome was identified a priori.

ELIGIBILITY:
Inclusion Criteria:

* SPIN Cohort patients must have a systemic sclerosis (SSc) diagnosis based on 2013 American College of Rheumatology/European League Against Rheumatism criteria confirmed by a SPIN physician, be ≥18 years old, be able to give informed consent, and be fluent in English, French or Spanish.
* For the feasibility trial, eligible patients must be able to use the online intervention in English, and have low disease management self-efficacy (Self-Efficacy for Managing Chronic Disease (SEMCD) ≤ 7).
* For the full-scale trial, eligible patients must be able to use the online intervention in English or French, and have low disease management self-efficacy (Self-Efficacy for Managing Chronic Disease (SEMCD) ≤ 7).

Exclusion Criteria:

* Patients not able to access or respond to questionnaires via the internet are excluded.
* Participants who are currently participating in another SPIN intervention trial and have not yet completed their final assessment measures will be excluded.
* French and Spanish speaking participants will be excluded from the feasibility trial.
* Spanish speaking participants will be excluded from the full-scale trial.
* Participants in the feasibility trial will be excluded in the full-scale trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease (SEMCD) Scale | 3 months
  The 6-item SEMCD Scale measures self-efficacy among patients with chronic medical conditions by asking them to rate their confidence that they can perform certain tasks related to managing their disease. Items are rated on a numerical scale ranging from 1 (not confident at all) to 10 (totally confident). The score for the scale is the mean of all item scores, with higher scores reflecting greater self-efficacy.

SECONDARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease (SEMCD) Scale | 6 months
  The 6-item SEMCD Scale measures self-efficacy among patients with chronic medical conditions by asking them to rate their confidence that they can perform certain tasks related to managing their disease. Items are rated on a numerical scale ranging from 1 (not confident at all) to 10 (totally confident). The score for the scale is the mean of all item scores, with higher scores reflecting greater self-efficacy.
Patient Activation Measure (PAM-13) | 3 months, 6 months
  Patient activation is determined by the extent to which patients effectively engage with and manage their own health. The 13-item patient activation measure (PAM-13) includes statements related to participants' attitudes and perspectives about their health, with four possible responses ranging from (1) strongly disagree to (4) strongly agree, with an additional "Not applicable" option. Using calibration tables (accessed with a purchased license), participants' responses are converted into raw scores ranging from 0-100, with higher scores indicating higher activation. Raw scores are sorted into four activation levels, with higher levels characterizing higher patient activation: (level 1) disengaged and overwhelmed, (level 2) becoming aware but still struggling, (level 3) taking action, (level 4) maintain behaviours and pushing further.
Social Appearance Anxiety Scale (SAAS) | 3 months, 6 months
  Changes in appearance that can occur due to systematic sclerosis (SSc) can cause a fear of social situations in which one's appearance is evaluated, or social appearance anxiety. The SAAS consists of 16 items that measure patients' self-reported anxiety related to situations where one's appearance will be evaluated, with response options ranging from 1 ("Not at all") to 5 ("Extremely"). To calculate total scores the first item ("I feel comfortable with the way I appear to others") is reverse-coded, all items are summed, and total scores range from 16-80, with higher scores indicating greater anxiety.
Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 | 3 months, 6 months
  Measures 8 domains of health status with 4 items for each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference) plus a single item for pain intensity. Items are scored on a 5-point scale (range 1-5), with different response options for different domains, and the single pain intensity item is measured on an 11-point rating scale. Higher scores represent more of the domain being measured
Participant Satisfaction: SPIN-SELF Program | 3 months
  Participant satisfaction with the SPIN-SELF Program will be evaluated with the Client Satisfaction Questionnaire-8 (CSQ-8), a standardized survey that is used to assess satisfaction with health services. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with total scores ranging from 8 to 32 and higher scores indicating greater satisfaction with the program. This measure will only be administered to participants in the intervention arm.
Patient Education Assessment Tool (PEMAT) | 3 months
  Participants will also be asked to answer open-ended questions about their experiences taking part in the SPIN-SELF Program, including difficulties, positive elements and other salient issues. Data collection will be done using an adapted version of the Patient Education Assessment Tool (PEMAT) questionnaire.
Usage of the SPIN-SELF Program internet modules | 3 months
  Usage of the SPIN-SELF Program internet modules among participants in the intervention arm will be examined via intervention usage data that will be collected automatically. These data will provide detailed information on the number of logins, number of modules accessed, goals set, and time spent on each webpage.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after the collection of the primary outcome
Access Criteria: Approval of proposed purpose for data access

REFERENCES:
- [Derived] Nordlund J, Henry RS, Kwakkenbos L, Carrier ME, Levis B, Nielson WR, Bartlett SJ, Dyas L, Tao L, Fedoruk C, Nielsen K, Hudson M, Pope J, Frech T, Gholizadeh S, Johnson SR, Piotrowski P, Jewett LR, Gordon J, Chung L, Bilsker D, Levis AW, Turner KA, Cumin J, Welling J, Fortune C, Leite C, Gottesman K, Sauve M, Rodriguez-Reyna TS, Larche M, van Breda W, Suarez-Almazor ME, Wurz A, Culos-Reed N, Malcarne VL, Mayes MD, Boutron I, Mouthon L, Benedetti A, Thombs BD; SPIN Investigators. The Scleroderma Patient-centered Intervention Network Self-Management (SPIN-SELF) Program: protocol for a two-arm parallel partially nested randomized controlled feasibility trial with progression to full-scale trial. Trials. 2021 Nov 27;22(1):856. doi: 10.1186/s13063-021-05827-z. PMID 34838105